CLINICAL TRIAL: NCT00553709
Title: The Role of Transcutaneous Nicotine in the Prevention of Postoperative Nausea and Vomiting in Non-smokers
Brief Title: Study of Nicotine for the Prevention of PONV
Acronym: NicoPONV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected difficult recruitment. Study drug expired
Sponsor: University Hospital, Geneva (Other)
Responsible Party: University Hospital, Geneva, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006DR3327; APSIC 04-010
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea; vomiting; retching; emesis; surgery; anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine patch (Experimental): Nicotinell® Patch 10 cm2, containing 17.5 mg of nicotine, with an average delivery rate of 7 mg of nicotine per 24 hours (= TTS 10)
  Interventions: Drug: Nicotine
- Placebo patch (Placebo Comparator): Placebo patch 10 cm2
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Nicotinell® Patch 10 cm2, containing 17.5 mg of nicotine, with an average delivery rate of 7 mg of nicotine per 24 hours (= TTS 10)

SUMMARY:
The purpose of this study is to determine whether nicotine is effective in the prevention of nausea and vomiting in non-smokers undergoing surgery

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 years)
* ASA I-II, non-smokers (or ex-smokers who have not been smoking for more than 2 years)
* Undergoing elective surgery (ENT, abdominal, urological, gynaecological); and
* Consenting to take part in the study will be included.

Exclusion Criteria:

* Smokers (cigarette, pipe, cigar)
* Patients undergoing nicotine replacement therapy
* Prolonged postoperative intubation
* Postoperative nasogastric tube

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Prevention of PONV | 48 hours postoperatively

SECONDARY OUTCOMES:
Adverse effects that may be related to the nicotine patch, for instance, local skin reaction. | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Tramèr, MD, DPhil, Study Chair — University Hospital, Geneva; Daniel Bertrand, PhD, Study Chair — Medical Faculty, Geneva University
Locations (1):
- Division of Anesthesiology, Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland